CLINICAL TRIAL: NCT04988893
Title: Quality of Recovery Scores in Parturients With Obesity: A Prospective Observational Cohort Study
Brief Title: Quality of Recovery Scores in Parturients With Obesity
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Other Study IDs: 11292
Record Dates: First submitted 2021-07-13; First posted 2021-08-04 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Quality of Recovery; Post Operative Pain
Keywords: Cesarean Section; Parturients; Morbid Obesity
MeSH Terms: conditions — Pain, Postoperative; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parturients with Normal Weight: Parturients undergoing elective caesarean delivery with a BMI <30 (control group)
- Parturients with Morbid Obesity: Parturients undergoing elective caesarean delivery with a BMI >40 (Study Group)

SUMMARY:
The prevalence of obesity has increased dramatically recently. Obesity is a pro-inflammatory state which leads to chronic low grade inflammation having different systemic effects. This may make obesity an independent risk factor for severe acute postoperative pain. No prospective studies have been conducted to specifically evaluate the quality of recovery after caesarean delivery for women with morbid obesity when compared to non-obese parturients. In addition, while there is biological plausibility to infer worse pain scores in parturients with obesity, the magnitude of this difference is unknown and information guiding adjustments in pain management are lacking.

DETAILED DESCRIPTION:
The prevalence of obesity has increased dramatically over the recent past in both developed and developing countries.

Obesity is a pro-inflammatory state which leads to chronic low grade inflammation. It has been well studied that this very inflammation and oxidative stress is responsible for cardiovascular pathologies seen in these patients. As a result, the post-operative period is characterized by a phase of prolonged systemic inflammatory response, which makes obesity an independent risk factor for severe acute pain. As a matter of fact, an extreme rise in IL-6 in patients with obesity has been demonstrated post-operatively.

In addition, adipose tissue acts as an endocrine organ by releasing a number of other pro-inflammatory proteins. Cytokines are known to promote various metabolic, hemodynamic and immunologic changes post-surgery, and in the setting of exaggerated inflammatory response can lead to increased pain and hemodynamic instability.

Very few studies have evaluated the recovery experience of patients with obesity in the acute postoperative period. Patients with obesity undergoing general abdominal surgery have been shown to have worse surgical outcomes, increased complication rates, and increased analgesic requirements.7 However, in spine surgery, there have been conflicting evidence supporting a difference in pain scores in patients with obesity. Despite there being no clear guidelines on post-operative pain control between these two groups, providers reported prescribing less opioid analgesics post-operatively to patients with obesity when compared to patients not suffering from this condition.

The Obstetric Quality of Recovery Score (ObsQoR) was initially developed and validated as a measure of patient reported outcome after caesarean delivery. It started as an 11-item questionnaire (ObsQoR-11), which was further simplified to 10-items (ObsQoR-10) following patient feedback where moderate and severe pain questions were combined into a single item. This tool measures pain, nausea or vomiting, dizziness, shivering, comfort, mobility, ability to hold and feed the baby, personal hygiene maintenance, and feeling in control, to provide a global inpatient postpartum quality of recovery score out of 100. A systematic review assessing measurement properties of available patient-reported outcome measures using COSMIN (COnsensus-based Standards for the selection of health Measurement INstruments) methodology, recommended ObsQoR as the best available instrument to measure functional recovery following caesarean delivery.

No prospective studies have been conducted to specifically evaluate the quality of recovery after caesarean delivery for women with morbid obesity when compared to non-obese parturients. In addition, while there is biological plausibility to infer worse pain scores in parturients with obesity, the magnitude of this difference is unknown and information guiding adjustments in pain management are lacking.

The investigators hypothesize that parturients with Class 3 obesity experience impaired quality of recovery scores after elective cesarean delivery as measured by the ObsQoR-10 when compared to non-obese parturients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Term pregnancy (> 37 weeks gestational age)
* Elective caesarean delivery
* BMI >40 (Study Group) or BMI <30 (Control Group)
* ASA<=3

Exclusion Criteria:

* Chronic pain
* History of opioid use during pregnancy.
* History of substance abuse disorder during pregnancy.
* Contraindication to neuraxial opioids, acetaminophen and/or NSAIDs
* Language barrier
* Allergy to Opioids or NSAIDS
* Intra-operative conversion to general anesthesia
* Maternal Admission to ICU.
* Neonatal admission to NICU.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects currently pregnant undergoing elective cesarean delivery
Study Population: Pregnant women meeting inclusion and exclusion criteria who are scheduled to have their Caesarean Section at Victoria Hospital, London Health Sciences Centre will be consented for participation in the study. Patients will be recruited from obstetrical and preadmission clinics at LHSC Victoria Hospital, as well as at admission for Caesarean Section to the Obstetrical Care Unit. Patients will be recruited only when inclusion criteria are fulfilled, in the absence of exclusion criteria, and after informed consent has been obtained.
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-03-18 (Actual)

PRIMARY OUTCOMES:
Difference in Obstetric Quality of Recovery Score (ObsQoR-10) | 24 hours post cesarean delivery
  10-item questionnaire applied to subjects 24 hours after spinal anesthesia. Measured in a 0-100 scale where 0=poor recovery and 100=perfect recovery

SECONDARY OUTCOMES:
Difference in Average Numeric Rating Score (0-10 , where 0=no pain and 10= maximum pain) at specific time points in the first 24 hours | Immediately after surgery (in PACU) and every 4 hours up to 24 hours after surgery
  This is defined as the between- group difference in the mean pain scores on a 0-10 Numeric Rating Scale, as assessed by one of the investigators immediately after surgery (in the Post-Anaesthesia Care Unit) and every 4 hours up to 24 hours after surgery
Opioid Consumption in the first 24 hours | 24 hours post cesarean delivery
  Between-group difference in the total amount of Oral Morphine Equivalents consumed in the first 24 hours after surgery.
Total Inpatient Opioid Consumption | up to 1 week post operatively
  Between-group difference in the total amount of Oral Morphine Equivalents consumed during hospital stay.
Time-to-first oral opioid analgesic request | Measured in hours from the time of cesarean delivery until patient request for prescribed oral opioid analgesia, up to 24 hours from the spinal anesthetic
  This is defined as the length of time between cesarean delivery and the first time the subject requested additional opioid analgesia
Respiratory Depression | In post-anesthesia care unit (PACU), and every 4 hours up to 24 hours after surgery
  This is defined as respiratory rate<8 breaths/minute, need for naloxone or need for clinical intervention.
Nausea and/or Vomiting that required treatment | Absolute number of treatments required in the 24-hour time frame
  Nausea/Vomiting episodes that required pharmacological treatment in the first 24 hours post operatively
Pruritus that required treatment | Absolute number of treatments required in the 24-hour time frame.
  Pruritus episodes that required pharmacological treatment in the first 24 hours post operatively
Breastfeeding | 24 hours post cesarean delivery
  Mother breastfeeding at 24 hours: Yes or No
Time to fist mobilization | Measured in hours from the time of cesarean delivery until patient first mobilizes post operatively, up to 48 hours post operatively.
  Time to fist mobilization (standing and walking independently): measured in hours
Time to first oral intake | Measured in hours from the time of cesarean delivery, up to 48 hours post operatively
  Time to first oral intake (non-clear fluids): measured in hours
Length of hospital stay | Measured in hours from the time of cesarean, up to to 1 month post operatively (average 48-72 hours)
  Length of hospital stay: measured in hours.
Unplanned Readmission Rates | 6 weeks post op
  Unplanned Readmission Rates prior to 6-week follow up appointment: Yes or No and reason for readmission

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Sebbag, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent HK, Taylor AG. Biomarkers and potential mechanisms of obesity-induced oxidant stress in humans. Int J Obes (Lond). 2006 Mar;30(3):400-18. doi: 10.1038/sj.ijo.0803177. PMID 16302012
- [Background] Musaad S, Haynes EN. Biomarkers of obesity and subsequent cardiovascular events. Epidemiol Rev. 2007;29:98-114. doi: 10.1093/epirev/mxm005. Epub 2007 May 10. PMID 17494057
- [Background] Mei W, Seeling M, Franck M, Radtke F, Brantner B, Wernecke KD, Spies C. Independent risk factors for postoperative pain in need of intervention early after awakening from general anaesthesia. Eur J Pain. 2010 Feb;14(2):149.e1-7. doi: 10.1016/j.ejpain.2009.03.009. Epub 2009 May 6. PMID 19423369
- [Background] Gletsu N, Lin E, Zhu JL, Khaitan L, Ramshaw BJ, Farmer PK, Ziegler TR, Papanicolaou DA, Smith CD. Increased plasma interleukin 6 concentrations and exaggerated adipose tissue interleukin 6 content in severely obese patients after operative trauma. Surgery. 2006 Jul;140(1):50-7. doi: 10.1016/j.surg.2006.01.018. PMID 16857442
- [Background] Galic S, Oakhill JS, Steinberg GR. Adipose tissue as an endocrine organ. Mol Cell Endocrinol. 2010 Mar 25;316(2):129-39. doi: 10.1016/j.mce.2009.08.018. Epub 2009 Aug 31. PMID 19723556
- [Background] Kim MG, Yook JH, Kim KC, Kim TH, Kim HS, Kim BS, Kim BS. Influence of obesity on early surgical outcomes of laparoscopic-assisted gastrectomy in gastric cancer. Surg Laparosc Endosc Percutan Tech. 2011 Jun;21(3):151-4. doi: 10.1097/SLE.0b013e318219a57d. PMID 21654297
- [Background] Elsamadicy AA, Camara-Quintana J, Kundishora AJ, Lee M, Freedman IG, Long A, Qureshi T, Laurans M, Tomak P, Karikari IO. Reduced Impact of Obesity on Short-Term Surgical Outcomes, Patient-Reported Pain Scores, and 30-Day Readmission Rates After Complex Spinal Fusion (>/=7 Levels) for Adult Deformity Correction. World Neurosurg. 2019 Jul;127:e108-e113. doi: 10.1016/j.wneu.2019.02.165. Epub 2019 Mar 12. PMID 30876992
- [Background] Sorimachi Y, Neva MH, Vihtonen K, Kyrola K, Iizuka H, Takagishi K, Hakkinen A. Effect of Obesity and Being Overweight on Disability and Pain After Lumbar Fusion: An Analysis of 805 Patients. Spine (Phila Pa 1976). 2016 May;41(9):772-7. doi: 10.1097/BRS.0000000000001356. PMID 26656059
- [Background] Kruger MT, Naseri Y, Hohenhaus M, Hubbe U, Scholz C, Klingler JH. Impact of morbid obesity (BMI > 40 kg/m2) on complication rate and outcome following minimally invasive transforaminal lumbar interbody fusion (MIS TLIF). Clin Neurol Neurosurg. 2019 Mar;178:82-85. doi: 10.1016/j.clineuro.2019.02.004. Epub 2019 Feb 4. PMID 30739072
- [Background] Bui AH, Feldman DL, Brodman ML, Shamamian P, Kaleya RN, Rosenblatt MA, D'Angelo D, Somerville D, Mudiraj S, Kischak P, Leitman IM. Provider preferences for postoperative analgesia in obese and non-obese patients undergoing ambulatory surgery. J Pharm Policy Pract. 2018 May 17;11:9. doi: 10.1186/s40545-018-0138-x. eCollection 2018. PMID 29796284
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408
- [Background] Ciechanowicz S, Howle R, Heppolette C, Nakhjavani B, Carvalho B, Sultan P. Evaluation of the Obstetric Quality-of-Recovery score (ObsQoR-11) following non-elective caesarean delivery. Int J Obstet Anesth. 2019 Aug;39:51-59. doi: 10.1016/j.ijoa.2019.01.010. Epub 2019 Feb 2. PMID 30885691
- [Background] Sultan P, Kormendy F, Nishimura S, Carvalho B, Guo N, Papageorgiou C. Comparison of spontaneous versus operative vaginal delivery using Obstetric Quality of Recovery-10 (ObsQoR-10): An observational cohort study. J Clin Anesth. 2020 Aug;63:109781. doi: 10.1016/j.jclinane.2020.109781. Epub 2020 Mar 20. PMID 32203873
- [Background] Sharawi N, Klima L, Shah R, Blake L, Carvalho B, Sultan P. Evaluation of patient-reported outcome measures of functional recovery following caesarean section: a systematic review using the consensus-based standards for the selection of health measurement instruments (COSMIN) checklist. Anaesthesia. 2019 Nov;74(11):1439-1455. doi: 10.1111/anae.14807. Epub 2019 Aug 20. PMID 31429919
- [Background] Sultan P, Carvalho B. Postpartum recovery: what does it take to get back to a baseline? Curr Opin Obstet Gynecol. 2021 Apr 1;33(2):86-93. doi: 10.1097/GCO.0000000000000684. PMID 33395109
- See also: WHO. Fact Sheet: Obesity and overweight. 2006. — http://www.who.int/mediacentre/factsheets/fs311/en/
- See also: 17. Sealed Envelope Ltd. 2012. Power calculator for continuous outcome superiority trial — https://www.sealedenvelope.com/power/continuous-superiority/